CLINICAL TRIAL: NCT01352416
Title: Suppression Of Atrial Fibrillation With Ranolazine After Cardiac Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Corewell Health East (Other)
Collaborators: Beaumont Foundation of America (Other); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Ilana Kutinsky, Physician, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-101, IN-US-259-0114
Record Dates: First submitted 2011-05-04; First posted 2011-05-11 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery
Keywords: Suppress Atrial Fibrillation; heart bypass surgery; heart valve surgery
MeSH Terms: interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CABG surgery with Ranolazine (Active Comparator): Patient will undergo Coronary Artery Bypass Graft (open heart surgery) and will receive, Ranolazine 1000 mg (2-500mg tablets) twice daily. If intolerant to the study drug due to adverse effects,or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 500 mg (1-500mg tablet) twice daily.
  Interventions: Drug: Ranolazine
- CABG surgery with placebo (Placebo Comparator): Patient will undergo Coronary Artery Bypass Graft (open heart surgery) and will receive, Placebo 1000mg mg (2-500mg tablets)twice daily. If intolerant to the study drug due to adverse effects, or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 500mg (1-500mg tablet) twice daily.
  Interventions: Drug: Placebo
- Heart Valve surgery with Ranolazine (Active Comparator): Patient will undergo heart Valve surgery and will receive, Ranolazine1000mg (2-500 mg tablets) twice a day. If intolerant to the study drug due to adverse effects, or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 500 mg (1-500mg tablet) twice a day.
  Interventions: Drug: Ranolazine
- Heart Valve surgery with placebo (Placebo Comparator): Patient will undergo heart Valve surgery and will receive, Placebo 1000mg (2-500mg tablets) twice a day. If intolerant to the study drug due to adverse effects, or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 500mg (1-500mg tablet) twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine 1000mg (2-500mg tablets) twice daily. Starting 2 days prior to surgery, morning of surgery and up to 14 days post operative depending when the breathing tube is removed from the patient post operative. If intolerant to the study drug due to adverse effects or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 500mg (1-500mg tablet) twice daily
  Other Names: Ranexa
  Arms: CABG surgery with Ranolazine; Heart Valve surgery with Ranolazine
Drug: Placebo — Placebo 1000mg (2-500mg tablets) twice daily. Starting 2 days prior to surgery, morning of surgery and up to 14 days post operative depending when the breathing tube is removed from the patient post operative. If intolerant to the study drug due to adverse effects or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 500mg (1-500mg tablet) twice daily
  Other Names: inactive ingredients pill
  Arms: CABG surgery with placebo; Heart Valve surgery with placebo

SUMMARY:
The objective of this study is to show that ranolazine is a safe, viable and potent alternative for post-operative atrial fibrillation suppression in patients undergoing cardiac surgery

DETAILED DESCRIPTION:
A single center, double blind, prospective, randomized study for patients who are scheduled for elective cardiac surgery (Coronary Artery Bypass Graft [CABG], or valve or CABG and valve). All patients who meet criteria will be prospectively enrolled in a randomized fashion. Patients enrolled will be assigned to receive twice daily identical capsules containing either placebo or ranolazine. Study drug will be initiated 2 days before surgery. Patients will receive study drug throughout their hospitalization and be kept on it for a full 2 weeks post operatively. Patients will be seen in 2 weeks and receive a 30 day follow up contact visit.

ELIGIBILITY:
Inclusion Criteria:

* Indications for cardiac surgery (CABG, valve surgery or CABG and valve surgery, Able to provide informed consent.

Exclusion Criteria:

* Documented atrial fibrillation within the previous 3 months
* Ongoing therapy with suppressive antiarrhythmic drugs
* Patient currently on digoxin
* Emergent surgery
* Patient receiving hemodialysis
* Concomitant use of ketoconazole, diltiazem, verapamil
* Known tolerance or hypersensitivity to ranolazine
* Pregnant individuals
* MAZE procedure (is a surgical ablation to treat atrial fibrillation) performed during concurrent cardiac surgery

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Kutinsky, DO, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started October 2010 and completed November 2012
Groups:
- Ranolazine and Patients Having CABG Surgery; Ranolazine With Patients Having Non CABG Heart Surgery: 500 mg tab, 2 pills twice a day. If intolerant to the study drug due to adverse effects,or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 500 mg, 1 pill twice daily.
  Atrial fibrillation : Once patient is in atrial fibrillation, the study drug is still continued. Patients will also be treated with standard drug therapy that their doctor chooses
- Sugar Pill and Patients Having CABG Surgery; Sugar Pills and Patients Having Non CABG Heart Surgery: 2 pills twice a day. If intolerant to the study drug due to adverse effects, or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 1 pill twice daily.
  Atrial fibrillation : Once the patient goes into atrial fibrillation, the study drug is still continued. Patient will also be treated with standard drug therapy that their doctor chooses
Period: Overall Study
Arm/Group | Ranolazine and Patients Having CABG Surgery | Sugar Pill and Patients Having CABG Surgery | Ranolazine With Patients Having Non CABG Heart Surgery | Sugar Pills and Patients Having Non CABG Heart Surgery
Started | 4 | 7 | 2 | 2
Completed | 3 | 5 | 0 | 1
Not Completed | 1 | 2 | 2 | 1
Not completed — Physician Decision | 1 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Subjects scheduled/undergoing cardiac surgery.
Groups:
- Ranolazine and Patients Having Heart Bypass Surgery; Ranolazine and Patients Having Non Heart Bypass Surgery: 500 mg tab, 2 pills twice a day. If intolerant to the study drug due to adverse effects,or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 500 mg, 1 pill twice daily.
  Atrial fibrillation : Once patient is in atrial fibrillation, the study drug is still continued. Patients will also be treated with standard drug therapy that their doctor chooses
- Placebo Pill and Patients Having Heart Bypass Surgery; Placebo Pill and Patients Having Non Heart Bypass Surgery: 2 pills twice a day. If intolerant to the study drug due to adverse effects,or the patient is started on diltiazem or verapamil post operative then the dose will be reduced to 500 mg, 1 pill twice daily.
  Atrial fibrillation : Once patient is in atrial fibrillation, the study drug is still continued. Patients will also be treated with standard drug therapy that their doctor chooses
- Total: Total of all reporting groups
Arm/Group | Ranolazine and Patients Having Heart Bypass Surgery | Placebo Pill and Patients Having Heart Bypass Surgery | Ranolazine and Patients Having Non Heart Bypass Surgery | Placebo Pill and Patients Having Non Heart Bypass Surgery | Total
Number analyzed (Participants) | 4 | 7 | 2 | 2 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 1 | 1 | 7
  >=65 years | 3 | 3 | 1 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (4.6) | 63.4 (9.9) | 48.0 (25.5) | 71.0 (9.9) | 63.4 (12.1)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 4 | 7 | 2 | 2 | 15
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 2 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Any Episode of Post Operative Atrial Fibrillation Longer Than 6 Hours Duration Occurring During the Study Period.
Description: Freedom from any episode of post operative Atrial Fibrillation (AF) longer than 6 hours duration occurring during the study period. To document post operative atrial fibrillation.
Time Frame: The time between the completion of the operation and hospital discharge or 14 days post operative if the hospitalzation is prolonged
Population: Study was prematurely terminated. Data for this Outcome Measure were not collected
Groups:
- Ranolazine With Coronary Artery Bypass Graft (CABG): Ranolazine 500 mg 2 pills twice a day with Coronary Artery Bypass Graft (CABG)
- Placebo With CABG: Placebo 2 pills twice daily with CABG
- Ranolazine Without CABG: Ranolazine 500 mg 2 pills twice daily without CABG
- Placebo Without CABG: Placebo 2 pills twice daily without CABG
Arm/Group | Ranolazine With Coronary Artery Bypass Graft (CABG) | Placebo With CABG | Ranolazine Without CABG | Placebo Without CABG
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All unexpected Adverse Events will be reported for the duration of the study. Subjects were followed and monitored for 30 days (duration of participation). Adverse events were collected for 2 years. Study was prematurely terminated.
Arm/Group | Ranolazine and Patients Having Heart Bypass Surgery | Placebo Pill and Patients Having Heart Bypass Surgery | Ranolazine and Patients Having Non Heart Bypass Surgery | Placebo Pill and Patients Having Non Heart Bypass Surgery
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Early termination due to lack of enrollment. 15 pts enrolled, 6 withdrawn due breathing tube not removed by 10 pm day of surgery. 1 withdrawn after day 3 as he was in afib and placed on amio. All pts were male.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No